CLINICAL TRIAL: NCT06620159
Title: Lymphocyte to Procalcitonin Ratio: A New Predictor of Prognosis and Mortality in Covid
Brief Title: Lymphocyte to Procalcitonin Ratio in Covid-19 Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Teslime Eryavuz Şengül, medical doctor, Suleyman Demirel University
Other Study IDs: SuleymanDU-MED-TEŞ-02
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid19(+): Covid19 patients with a positive PCR test

SUMMARY:
The lymphocyte/CRP ratio has been studied many times in covid-19 patients and has been proven to be an indicator of mortality as well as poor prognosis. In this study, the role of the lymphocyte/procalcitonin ratio in predicting the hospitalization status of patients, detection of findings on CT, need for mechanical ventilation, mortality and survival is aimed to be determined. The lymphocyte/procalcitonin ratio was found to be the strongest predictor of mortality and poor prognosis, especially in patients over 65 years of age.

DETAILED DESCRIPTION:
The lymphocyte/CRP ratio has been studied many times in covid-19 patients and has been proven to be an indicator of mortality as well as poor prognosis. In this study, the role of the lymphocyte/procalcitonin ratio in predicting the hospitalization status of patients, detection of findings on CT, need for mechanical ventilation, mortality and survival is aimed to be determined. The lymphocyte/procalcitonin ratio was found to be the strongest predictor of mortality and poor prognosis, especially in patients over 65 years of age. The auc value, PPV and specificity of the lymphocyte/procalcitonin ratio were higher than the lymphocyte/CRP ratio.

ELIGIBILITY:
Inclusion Criteria:

* Covid19 PCR test positive

Exclusion Criteria:

* Pregnancy Under 18 years old

Ages: 23 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who applied to suleyman demirel university emergency department and diagnosed with covid 19 by PCR
Sampling Method: Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
outcome | 30 days
  The relationship between lymphocyte/procalcitonin ratio and 30-day mortality was analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Furkan Ç Oğuzlar, asst. prof., Principal Investigator — suleyman demirel university faculty of medicine
Locations (1):
- Süleyman demirel üniversitesi tıp fakültesi, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No